CLINICAL TRIAL: NCT02766595
Title: Hyperventilation During Routine EEG in Children: the Impact of Body Position - Sitting vs Supine- on the Yield of the Procedure in Provoking Absence Seizures
Brief Title: Does Body Positioning Affect the Yield of Hyperventilation in Routine Pediatric Electroencephalography - EEG Studies?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0257-15-MMC
Record Dates: First submitted 2016-03-10; First posted 2016-05-10 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-03

CONDITIONS: Epilepsy, Absence
MeSH Terms: conditions — Epilepsy, Absence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hyperventilation (Other): Non-drug: performing hyperventilation while sitting up during routine EEG
  Interventions: Other: hyperventilation while sitting up during routine EEG

INTERVENTIONS:
Other: hyperventilation while sitting up during routine EEG — Child will be asked to perform hyperventilation while lying down as well as while sitting up

SUMMARY:
Children referred for routine EEG studies for suspected absence seizures will be asked, upon caregiver's informed consent, to perform 3 minutes of hyperventilation both in the supine position and while sitting up. We aim to demonstrate that hyperventilation is more effective in eliciting absence seizures in a sitting position than while lying down.

DETAILED DESCRIPTION:
Hyperventilation is a very effective means of eliciting absence seizures in children with absence epilepsy. Worldwide EEG protocols for routine EEG recording include 3 minutes of hyperventilation. The whole EEG recording, including hyperventilation, is performed with the child lying down on a bed/coach. Our clinical experience suggests that the body position may affect the yield of hyperventilation in provoking the absence event. That is, hyperventilation may be more effective when the child is sitting up, Therefore, children referred for a routine EEG for suspected absence seizures will add 3 minutes of hyperventilation on a sitting position to the routine 3 minutes of supine hyperventilation. At least 5 minutes of rest will be allotted between both procedures.

Patients' caregivers will sign an informed consent form. Patients will randomly be divided into 2 groups: one group will first perform supine hyperventilation followed by sitting hyperventilation; the second group will perform hyperventilation in the opposite order, ie, first sitting up and then in supine position.

ELIGIBILITY:
Inclusion Criteria:

* Children referred for a routine EEG for suspected absence epilepsy

Exclusion Criteria:

* Patients unable to perform hyperventilation
* Children previously diagnosed with absence epilepsy
* Children receiving antiepileptic drugs

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-01 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Differences in elapsed time (in seconds) to onset of absence seizure between lying supine and sitting up during hyperventilation in routine EEG. | 6 months
  patients to be divided into 3 groups: Response A: occurrence of absence within 0-60 seconds; response B: within 60 - 120 seconds; response C: no occurrence of absence.

SECONDARY OUTCOMES:
Influence of order of performing hyperventilation, first supine and then sitting up, or vice-versa, on the time (in seconds) to occurrence of ansence seizures | 6 months
  Response A: 0 - 60 secs; response B: 60 - 120 seconds; response C: no occurrence of absence

IPD SHARING:
Plan to Share IPD: No